CLINICAL TRIAL: NCT02678494
Title: Home Based Brain-Train Treatment of Central Neuropathic Pain Following Spinal Cord Injury
Brief Title: Brain-Train Home Based Pain Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN15NE124
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2017-08

CONDITIONS: Neuropathic Pain
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurofeedback training (Experimental): Neurofeedback training: self-administered at home for 3 months. 3-5 sessions per week initially, then at least once a week. Each session consists of 5-6 blocks of 5 minute training.
  Interventions: Other: Neurofeedback training

INTERVENTIONS:
Other: Neurofeedback training

SUMMARY:
A study examining the effectiveness of neurofeedback therapy for the treatment of Central Neuropathic Pain (CNP), in patients with a Spinal Cord Injury, using a small user-friendly device which can be operated by patients at home.

DETAILED DESCRIPTION:
Spinal Cord Injury (SCI) affects a person's ability to move and feel sensation from the body. SCI is also an indirect cause of a persistent pain, called Central Neuropathic Pain (CNP). This pain typically develops several months after the injury.

In 30% to 40% of SCI patients, severe CNP affects their everyday living including sleep and mood. Medical treatment of CNP is moderately effective and costly, both to the patient and to the health care system.

In a previous study, some characteristic 'signatures' of brain waves that are related to CNP were defined. Based on this, a novel treatment for CNP based on neurofeedback was developed and clinically tested on five SCI patients. Electroencephalograph (EEG) was used to record patients' brain waves and shown to patients on a computer screen in a simple graphical form (e.g. bars). Patients were trained to change their brain activity at will and, as a consequence, their pain was reduced. Costly laboratory devices were used and once the study was over, an adequate alternative could not be offered to patients.

In this study, a cheap, portable, wireless and user friendly, Conformité Européenne (CE) marked EEG device will be used to train 10 patients to self-administer the therapy in the comfort of their homes. Participants will be given initial training to use the equipment then will be asked to use the system at home for 3 months - initially, 3-5 times a week then, if/when pain subsides, at least once a week or as required.

The primary purpose of the study is to determine whether a portable system for neuromodulation is a useful tool for administering therapy for pain (intensity of pain will be measured by the visual numerical scale (VNS)).

The secondary purpose of the study is a quantitative analysis of changes in the brain activity due to therapy, as measured by EEG; patients' perspective of the home based neuro-therapy (assessed by questionnaires and one-to-one, semi-structured interviews).

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal vision
* no history of brain disease or injury
* incomplete/complete injury at level C5 to T12
* central neuropathic pain (below the level of injury)
* intensity of pain 4 or above (VNS)
* stable medication regime (expected not to change during the period of the study), responding to some extent to CNP medication treatment
* patient or caregiver minimum computer literacy (owning a computer, laptop, tablet, ipad etc)

Exclusion Criteria:

* chronic or acute muscular or visceral pain larger than 4 VNS
* epilepsy
* diagnosed mental health problems
* active intervention of pain team (changing existing treatments)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06-09 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline and 3 months
  Change in intensity of pain as measured by the Visual Numerical Scale

SECONDARY OUTCOMES:
Brain activity | Baseline and 3 months
  Change in brain activity as measured by EEG
Patients' perspective of home-based neuro-therapy training | 3 months
  Qualitative assessment of patient's perspective of treatment as assessed by questionnaire and one-to-one semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Vuckovic, Dipl Ing MSc PhD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom